CLINICAL TRIAL: NCT03362047
Title: Untersuchung Des Einflusses PAH-spezifischer Medikation Auf Die rechtsventrikuläre Funktion Bei Patienten Mit Pulmonaler Arterieller Hypertonie (PAH) Unter Basalen Bedingungen
Brief Title: (RIGHT HEART III Study - Right Ventricular Hemodynamic Evaluation and Response to Treatment)
Acronym: RightHeartIII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 250774; 2015-002835-17 (EudraCT Number)
Record Dates: First submitted 2017-11-22; First posted 2017-12-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: Multicentre, randomized, prospective, open pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Riciguat Group (Experimental): 15 PAH patients will be administered Riciguat according to standard of care. RV function will be evaluated 90 mintutes after first medication intake and 12 weeks after first medication intake.
  Interventions: Drug: Riciguat Group
- Macitentan Group (Experimental): 15 PAH patients will be administered Macitentan according to standard of care. RV function will be evaluated 90 mintutes after first medication intake and 12 weeks after first medication intake.
  Interventions: Drug: Macitentan Group

INTERVENTIONS:
Drug: Riciguat Group — Patients will be administered 12 weeks Riciguat
  Arms: Riciguat Group
Drug: Macitentan Group — Patients will be administered 12 weeks Macitentan
  Arms: Macitentan Group

SUMMARY:
Pilot study to determine the therapeutic effect of two prarallel groups treated with either Riciguat or Macitentan, evaluated by the change in systolic and diastolic RV function within 12 weeks after first drug intake in order to plan a larger Phase II study.

DETAILED DESCRIPTION:
In this multi-center, randomized, open pilot study the therapeutic effect of two prarallel groups treated with either Riciguat or Macitentan shall be determined by evaluating the change in systolic and diastolic RV function within 12 weeks after first drug intake in order to plan a larger Phase II study.The method used to determine the RV function will be the "Conductance Method".

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients, 18 years ≤ age ≤ 85 years
* Diagnosis of Pulmonary Hypertension Group 1 according to Nizza Definition (PAH) confirmed by invasive methods, WHO functional class II and III
* Existing clinical need to repeat a right ventricular catheter examination (as recommended by the current "Kölner Konsensuskonferenz")
* Ability to understand study goals and agree to study participation
* Hemodynamic criteria of ventricular catheter examination:

  * Pulmonary vascular resistance (PVR)> 240 dyn x sec x cm-5
  * Mean Pulmonary Arterial Pressure (mPAP) ≥ 25 mmHg
* Clinical need to receive treatment with a drug approved for the treatment of PAH for the first time
* Potentially fertile women must agree to use highly effective methods of contraception, either through abstinence or the use of at least two methods of contraception from the date of consent until one month after the end of the study. An effective pregnancy protection consists in the combination of a hormonal contraceptive (oral, injectable or implant) and a barrier method (condom or diaphragm with a vaginal spermicide)
* Written consent to the clinical trial

Exclusion Criteria:

Existing therapy with positive inotropic drugs such as Catecholamines (including norepinephrine, dobutamine, suprarenin)

* Pregnancy or breastfeeding
* General contraindication for examinations to be performed during the study
* Hypersensitivity to the active substances or to a constituent of the study medication (in particular lactose and soya)
* Simultaneous participation in another medical therapy study
* Simultaneous participation in another non-drug study that would preclude participation in this study
* Participation within one month after completing another therapy study
* Heavy liver function disorders
* Existing increase in liver aminotransferases (aspartate aminotransferase (AST) and / or alanine aminotransferase (ALT))> 3 × ULN
* Systolic blood pressure <95 mmHg
* Pulmonary hypertension associated with idiopathic interstitial pneumonia (PH-IIP)
* anemia (Hb <10 g / dl)
* Concomitant medication with potential interaction to macitentan and/or riociguat according to the IB
* Severe kidney dysfunction
* Severe hemoptysis
* History of bronchial artery embolization
* smoker

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
RV function | 12 weeks
  Evaluation of the therapeutic effect of both treatment groups as measured by the change in systolic and diastolic RV function within 12 weeks after starting medication to plan a larger Phase II study. Methods: RV Catheterisation and Conductance Catherterisation.

SECONDARY OUTCOMES:
recruitability | 12 months
  The feasible to include 30 patients within 12 months will be assessed by descripitve statistic
feasibility to set up a larger phase II study | 24 months
  The feasibility to set up a larger phase II study with this study setting and design will be assessed by descripitve statistic
RV contractility | 12 weeks
  Percent change in RV contractility (= end-systolic elastance, EES), RV, Methods: RV Catheterisation and Conductance Catherterisation.
Collection of Adverse Events | 12 weeks
  number of participants with adverse events (all) assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Werner Seeger, Prof, Principal Investigator — University Gießen
Locations (3):
- Germany (3):
  - Klinik III für Innere Medizin Herzzentrum der Universität zu Köln, Cologne
  - Abteilung Pneumologie und Intensivmedizin der Medizinischen Klinik II, Uniklinik Gießen und Marburg Standort Gießen, Giessen
  - Krankenhaus Neuwittelsbach, Innere Medizin II, München

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on request
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared after end of study without limitation
Access Criteria: e-mail to: Khodr.Tello@innere.med.uni-giessen.de

REFERENCES:
- [Background] McGoon MD, Benza RL, Escribano-Subias P, Jiang X, Miller DP, Peacock AJ, Pepke-Zaba J, Pulido T, Rich S, Rosenkranz S, Suissa S, Humbert M. Pulmonary arterial hypertension: epidemiology and registries. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D51-9. doi: 10.1016/j.jacc.2013.10.023. PMID 24355642
- [Background] Peacock AJ, Crawley S, McLure L, Blyth KG, Vizza CD, Poscia R, Francone M, Iacucci I, Olschewski H, Kovacs G, Vonk Noordegraaf A, Marcus JT, van de Veerdonk MC, Oosterveer FP. Changes in right ventricular function measured by cardiac magnetic resonance imaging in patients receiving pulmonary arterial hypertension-targeted therapy: the EURO-MR study. Circ Cardiovasc Imaging. 2014 Jan;7(1):107-14. doi: 10.1161/CIRCIMAGING.113.000629. Epub 2013 Oct 30. PMID 24173272
- [Background] Borgdorff MA, Bartelds B, Dickinson MG, Boersma B, Weij M, Zandvoort A, Sillje HH, Steendijk P, de Vroomen M, Berger RM. Sildenafil enhances systolic adaptation, but does not prevent diastolic dysfunction, in the pressure-loaded right ventricle. Eur J Heart Fail. 2012 Sep;14(9):1067-74. doi: 10.1093/eurjhf/hfs094. Epub 2012 Jun 22. PMID 22730335
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Respir J. 2015 Oct;46(4):903-75. doi: 10.1183/13993003.01032-2015. Epub 2015 Aug 29. PMID 26318161
- [Background] Ghofrani HA, Galie N, Grimminger F, Grunig E, Humbert M, Jing ZC, Keogh AM, Langleben D, Kilama MO, Fritsch A, Neuser D, Rubin LJ; PATENT-1 Study Group. Riociguat for the treatment of pulmonary arterial hypertension. N Engl J Med. 2013 Jul 25;369(4):330-40. doi: 10.1056/NEJMoa1209655. PMID 23883378
- [Background] Kojonazarov B, Sydykov A, Pullamsetti SS, Luitel H, Dahal BK, Kosanovic D, Tian X, Majewski M, Baumann C, Evans S, Phillips P, Fairman D, Davie N, Wayman C, Kilty I, Weissmann N, Grimminger F, Seeger W, Ghofrani HA, Schermuly RT. Effects of multikinase inhibitors on pressure overload-induced right ventricular remodeling. Int J Cardiol. 2013 Sep 10;167(6):2630-7. doi: 10.1016/j.ijcard.2012.06.129. Epub 2012 Jul 31. PMID 22854298
- [Background] Lang M, Kojonazarov B, Tian X, Kalymbetov A, Weissmann N, Grimminger F, Kretschmer A, Stasch JP, Seeger W, Ghofrani HA, Schermuly RT. The soluble guanylate cyclase stimulator riociguat ameliorates pulmonary hypertension induced by hypoxia and SU5416 in rats. PLoS One. 2012;7(8):e43433. doi: 10.1371/journal.pone.0043433. Epub 2012 Aug 17. PMID 22912874
- [Background] Brimioulle S, Wauthy P, Ewalenko P, Rondelet B, Vermeulen F, Kerbaul F, Naeije R. Single-beat estimation of right ventricular end-systolic pressure-volume relationship. Am J Physiol Heart Circ Physiol. 2003 May;284(5):H1625-30. doi: 10.1152/ajpheart.01023.2002. Epub 2003 Jan 16. PMID 12531727
- [Background] Herberg U, Gatzweiler E, Breuer T, Breuer J. Ventricular pressure-volume loops obtained by 3D real-time echocardiography and mini pressure wire-a feasibility study. Clin Res Cardiol. 2013 Jun;102(6):427-38. doi: 10.1007/s00392-013-0548-3. Epub 2013 Feb 9. PMID 23397593
- [Background] Wilkins MR, Paul GA, Strange JW, Tunariu N, Gin-Sing W, Banya WA, Westwood MA, Stefanidis A, Ng LL, Pennell DJ, Mohiaddin RH, Nihoyannopoulos P, Gibbs JS. Sildenafil versus Endothelin Receptor Antagonist for Pulmonary Hypertension (SERAPH) study. Am J Respir Crit Care Med. 2005 Jun 1;171(11):1292-7. doi: 10.1164/rccm.200410-1411OC. Epub 2005 Mar 4. PMID 15750042
- [Background] Nagendran J, Sutendra G, Paterson I, Champion HC, Webster L, Chiu B, Haromy A, Rebeyka IM, Ross DB, Michelakis ED. Endothelin axis is upregulated in human and rat right ventricular hypertrophy. Circ Res. 2013 Jan 18;112(2):347-54. doi: 10.1161/CIRCRESAHA.111.300448. Epub 2012 Dec 10. PMID 23233754
- [Background] Muller HH, Schafer H. A general statistical principle for changing a design any time during the course of a trial. Stat Med. 2004 Aug 30;23(16):2497-508. doi: 10.1002/sim.1852. PMID 15287080
- [Background] Timmesfeld N, Schafer H, Muller HH. Increasing the sample size during clinical trials with t-distributed test statistics without inflating the type I error rate. Stat Med. 2007 May 30;26(12):2449-64. doi: 10.1002/sim.2725. PMID 17080491
- [Background] Galie N, Barbera JA, Frost AE, Ghofrani HA, Hoeper MM, McLaughlin VV, Peacock AJ, Simonneau G, Vachiery JL, Grunig E, Oudiz RJ, Vonk-Noordegraaf A, White RJ, Blair C, Gillies H, Miller KL, Harris JH, Langley J, Rubin LJ; AMBITION Investigators. Initial Use of Ambrisentan plus Tadalafil in Pulmonary Arterial Hypertension. N Engl J Med. 2015 Aug 27;373(9):834-44. doi: 10.1056/NEJMoa1413687. PMID 26308684